CLINICAL TRIAL: NCT06600867
Title: Evaluation of a Method for Measuring Dental Mobility and Displacement Force in Incisors With Periodontal Support Loss
Brief Title: Method for Measuring Dental Mobility and Displacement Force
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Enilson Antonio Sallum, PhD, Head of the Periodontology Department, University of Campinas, Brazil
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 81525124.9.0000.5418
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Periodontal Disease; Mobility, Tooth
Keywords: Periodontal Disease; Tooth Mobility; Periodontal Attachment Loss
MeSH Terms: conditions — Periodontal Diseases; Tooth Mobility; Periodontal Attachment Loss

STUDY DESIGN:
Intervention Model Description: Descriptive interventional clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tooth Mobility Assessment (Experimental): Tooth Mobility and Applied Force Assessment
  Interventions: Diagnostic Test: Tooth mobility assessment

INTERVENTIONS:
Diagnostic Test: Tooth mobility assessment — The examiner, holding the instruments (two clinical mirror handles), will apply labial/lingual or labial/palatal displacement movements using the subjective technique, just as routinely done. Using the endodontic spacer and the stop, the deflection will be measured in millimeters. Subsequently, the examiner, with the instruments in hand (tensiometer and dynamometer), will apply labial/lingual and labial/palatal displacement movements, determining the force required to achieve the same displacement previously established by the subjective method (reference/limit of displacement).

SUMMARY:
This study aims to investigate the use of a new method for measuring tooth mobility, which includes control of force (gf) and labial/lingual/palatal displacement (mm) of upper and lower incisors with tooth mobility. It will take place during a single assessment session at the clinic of the Piracicaba Dental School (FOP-Unicamp), supervised by the research student Larissa Alexandra Fatinanzi and Prof. Dr. Enílson Antônio Sallum. The evaluation will be conducted in person during regular clinical appointments, without requiring additional travel or extended time beyond what is planned.

The research will be conducted over two different days of appointments, scheduled on the same day and time as regular clinical appointments, occupying 30 minutes to 1 hour each.

Day 1: A molding (copy of the tooth) will be performed. Based on this step, a customized instrument will be made (necessary for evaluating the tooth with mobility).

Customized Instrument: The materials used will include: acetate plate (similar to a teeth whitening tray); endodontic spacer (used in root canal treatment); tensiometer and dynamometer (used in orthodontics to measure force); and caliper (a device for measuring in millimeters).

Day 2: Evaluations will be conducted, including mobility (tooth with movement), periodontal parameters (examination of the gums and tooth support system), and completion of a questionnaire with basic questions relating daily life to the clinical situation (tooth with movement).

The assessment of dental mobility involves moving the tooth forward and backward, similar to routine clinical practice. The amount of tooth movement will be measured in millimeters using the customized instrument. Additionally, a tensiometer and dynamometer will be used to measure the force. The force applied by the instruments will not harm the tooth with mobility. Two sets of dental mobility tests will be performed, with a 1-minute interval between them. The instruments used pose no risk to oral tissues, are employed in dental treatments, and are non-invasive. All evaluations will be carried out on the same day of the appointment.

DETAILED DESCRIPTION:
This will be a descriptive study. The population will consist of 20 volunteers diagnosed with periodontitis in stages II, III, and IV and grades A, B, and C, meeting the following inclusion criteria: periodontal pockets ≥ 4 mm, anterior teeth (regions 13-23 and/or 33-43) with dental mobility (grades 1, 2, or 3) and periodontal attachment loss, aged 18 years or older.

Patient selection will initially be conducted through the electronic medical records of patients undergoing treatment at the Piracicaba Dental School - Unicamp clinic.

The research will be carried out at the Periodontology Clinic of the Piracicaba Dental School (FOP-Unicamp), and the participation of volunteers will occur during regular clinical appointments, under the responsibility of the masters student Larissa Alexandra Fatinanzi and supervision of Prof. Dr. Enílson Antônio Sallum.

The method for evaluating dental mobility will include the use of a custom-made mold tray (PET-G; Bio-Art Soluções Inteligentes) for each patient with adaptations for displacement readings, an adapted tensiometer (Morelli, Orthodontics), a dynamometer (Zeusan, Campinas), two mirror handles, an endodontic spacer with a stop, and a caliper (Mitutoyo, Illinois, USA). Initially, the participant will receive the Informed Consent Form (ICF), and upon acceptance, the creation of the mold tray will begin based on the plaster model. In the next step, periodontal parameters (PS, NIC, bone loss in mm and % bone loss), premature contacts, and occlusal interferences will be assessed, along with the OHIP-14 (Oral Health Impact Profile), followed by dental mobility assessment using the conventional method with subjective force (mirror handles). The subjective force will determine the tooth displacement in millimeters (mm), which will then be used to establish the necessary objective force (measured by the tensiometer/dynamometer) to achieve the same displacement. Mobility will be classified according to Lindhe and Nyman classification (1975).

The chosen and adapted instrument for this research is the Orthodontic Tensiometer (Morelli Orthodontics, Sorocaba/SP, Brazil), with the inclusion of the Dynamometer (Zeusan, Campinas/SP - Brazil) for comparison purposes. The force measurements are presented in gf (gram-force), ranging from 25gf to 250gf (tensiometer) and 12.5g to 300g. Both instruments in this study will allow for the objective assessment of the routinely used subjective force and its possible relationship with clinical levels of attachment, in order to understand the magnitude of the force needed to displace a dental element with periodontal disease. The dynamometer will serve as a comparison tool and to confirm the accuracy of the tensiometer.

For statistical analysis, the comparison between the two techniques will be applied within the same group of subjects. Each volunteer will serve as their own control, reducing inter-subject variability. Normal distribution will be tested using the Shapiro-Wilk test. Comparisons will be made using Students t-test.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Periodontitis Stage II, III, and IV (grades A, B,C) and with periodontal pockets ≥ 4 mm.
* Anterior teeth (13-23 and 33-43) with dental mobility (grade 1, 2, or 3).
* Aged ≥ 18 years.

Exclusion Criteria:

* Crossbite or end-to-end bite.
* Bruxism.
* Implants adjacent to the tooth with mobility.
* Extreme mobility.
* Occlusal trauma.
* Patients requiring prophylactic antibiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Tooth mobility: force control (gf) | immediately before the clinical assessment
  Assess the force (gf) needed for each patient/tooth to achieve the diagnostic displacement of lower and upper incisors exhibiting dental mobility
Tooth Mobility: labial-lingual/palatal displacement (mm) | immediately before the clinical assessment
  Assess the displacement of lower and upper incisors with dental mobility

SECONDARY OUTCOMES:
Compare two instruments for measuring force | At the end of the 3-months study
  adapted tensiometer versus dynamometer

OTHER OUTCOMES:
Quality of life (OHIP-14) questionnaire | At the end of the 3-months study
  Assess the impact of dental mobility on quality of life (OHIP-14)

CONTACTS AND LOCATIONS:
Overall Officials: Larissa A Fatinanzi, MsC, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Faculdade de Odontologia de Piracicaba, Universidade Estadual de Campinas, Piracicaba, São Paulo, Brazil